CLINICAL TRIAL: NCT02507570
Title: Open Label Phase Two Study of Enzalutamide With Concurrent Administration of Radium Ra 223 Dichloride in Castration-Resistant (Hormone-Refractory) Prostate Cancer Subjects With Symptomatic Bone Metastasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carolina Research Professionals, LLC (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRP-PCA-02 EnzaRadiCate
Record Dates: First submitted 2015-07-16; First posted 2015-07-24 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Prostate Carcinoma Metastatic to the Bone
MeSH Terms: interventions — enzalutamide; radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label (Experimental): Single arm study to evaluate safety and tolerability of Enzalutamide with concurrent administration of Radium ra 223 dichloride in subjects with symptomatic metastatic prostate cancer.
  Interventions: Drug: Enzalutamide; Radiation: Radium ra 223 dichloride

INTERVENTIONS:
Drug: Enzalutamide — used concomitantly
  Other Names: XTANDI and Xofigo
Radiation: Radium ra 223 dichloride

SUMMARY:
This is an open label study designed to examine the effects of Enzalutamide with concurrent administration of Radium Ra 223 dichloride in Castrate-Resistant (Hormone-Refractory) Prostate Cancer subjects with symptomatic bone metastases in both the pre- and post-chemotherapy setting.

DETAILED DESCRIPTION:
This is an open label study designed to examine the effects of Enzalutamide with concurrent administration of Radium Ra 223 dichloride in castrate resistant (hormone-refractory) prostate cancer subjects with symptomatic bone metastasis, in both the pre- and post- chemotherapy setting.

Radium Ra 223 dichloride is approved by the US Food and Drug Administration for this indication. Enzalutamide is US Food and Drug Administration approved for this indication.

Approximately 40 subjects will be enrolled to obtain 30 evaluable subjects. All subjects will receive Radium Ra 223 dichloride every 4 weeks for a total of 6 doses over 24 weeks and concurrent Enzalutamide for a minimum duration of 24 weeks. The sponsor will provide Enzalutamide after the End of Treatment visit until the last Long Term Follow Up visit has been completed. Subjects will continue to receive Enzalutamide as long as a positive response to therapy is demonstrated. Enzalutamide may be discontinued at any time per physician discretion.

Subjects will be evaluated 30 days after the last dose of Radium Ra 223 dichloride. Including screening, the total duration of the study is 32 weeks plus every 3 month follow up visits while subjects are receiving Enzalutamide.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects will conform to all of the inclusion criteria listed below:

1. Subject must be able to understand and be willing to sign the written Informed Consent Form. A signed IRB approved Informed Consent Form must be appropriately obtained prior to the conduct of any study-specific procedure.
2. Subject is willing and able to comply with the protocol, including all study visits and procedures.
3. Subject is a male, greater than 18 years at time of enrollment.
4. Life expectancy of at least 9 months.
5. Subject has histologically documented prostate cancer confirmed by a pathology report from a prostate biopsy or radical prostatectomy specimen.
6. Subject must:

1. have initiated a stable dose of daily Enzalutamide within 45 days of enrollment (Cycle 1/Week 1/ Day 1), or 2. plans to initiate a stable daily dose of Enzalutamide within 30 days of the first Radium Ra 223 dichloride treatment.

7. Subject must plan to receive all 6 Radium Ra 223 dichloride injections and daily oral doses of Enzalutamide during the study, per protocol.

8. Subject has a history of bone metastasis from prostate cancer as evidenced by imaging performed within 90 days of enrollment (Cycle 1/Week 1/Day 1) from one of the following:

1. Tc Bone Scan or 2. Sodium Fluoride PET/CT Scan

* If a bone scan is used, solitary lesions which could be contributed to causes other than prostate cancer must be confirmed with a second modality (i.e.: plain films, CT scan or MRI).

  9. Subject has Castrate Resistant Prostate Cancer, defined as having a rising PSA level and a testosterone level </= 50ng/dl (2.0 nM/L) while receiving androgen deprivation therapy (medical or surgical castration). Subject must also plan to receive androgen deprivation therapy throughout the study.
* PSA progression is defined as having at least 2 rising PSA levels taken at least 7 days apart, with the 2nd PSA being 2.0 ng/dl or greater.

  10. Subject has the presence of cancer related bone pain requiring treatment with analgesic medications (including but not limited to acetaminophen, NSAIDS, Cox-2 inhibitors, and narcotic opioids).

  11. Subject has an ECOG performance status of 0-2 at the screening and enrollment visits.

  12. Acceptable hematology and serum biochemistry screening values: White Blood Cell (WBC) >/= 3,000/mm3 Absolute Neutrophil Count (ANC) >1500/mm3 Platelet (PLT) count >100,000/mm3 Hemoglobin (HGB) > 10.0 g/dL (100g/L; 6.2 mmol/L Creatinine <1.5 ULN Total bilirubin level <1.5 X ULN Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5 X ULN albumin >25 g/L Baseline electrolytes within normal limits ( Sodium, potassium, chloride, calcium, phosphate, magnesium, LDH, γGT, urea, total protein)

  13. Normal Liver Function Tests (LFT) and normal Renal Function Tests (RFT) at the screening visit. If the subject has LFT's or RFT's greater than 2.5 times the upper limit of normal (ULN), Medical Monitor review, in conjunction with the subject's PI, will be required.

  14. Subjects receiving Anti-Resorptive medications, such as denosumab (XGEVA) and Zolendronic Acid (Zometa), must be on a stable dose for at least 90 days prior to enrollment (Cycle 1/Week 1/Day 1). Anti-resorptive medications may be not be added to the subject's regimen during the study. Anti-resorptive discontinuation will be allowed per Investigator discretion due to adverse events attributable to that medication.

  15. Subjects of childbearing potential must agree to use adequate contraception beginning at the enrollment until at least 30 days after the last dose of the study drugs. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate.

Exclusion Criteria:

Eligible subjects must not meet any of the exclusion criteria listed below:

1. Subject has known malignant pleural effusion, or known lung, liver or brain metastasis (lymph node only metastasis <6 cm in short-axis diameter is allowed).
2. Subject has a history of seizure or any condition that may predispose him to seizures (e.g. prior cortical stroke, significant brain trauma) at any time in the past, or a history of loss of consciousness or transient ischemic attack within 12 months of enrollment (Cycle 1/Week 1/Day 1).
3. Subject has received previous treatment with Enzalutamide for longer than 45 days prior to enrollment (Cycle 1/Week 1/Day 1), or any prior treatment with Radium Ra 223 dichloride.
4. Subject has a known medical contraindication to Enzalutamide or Radium Ra 223 dichloride.
5. Subject is not willing to initiate a stable dose of daily Enzalutamide within 45 days of enrollment (Cycle 1/Week1/Day 1), or does not plan to initiate a stable daily dose of Enzalutamide within 30 days of the first Radium Ra 223 dichloride treatment (Cycle 1/Week 1/Day 1).
6. Subject does not plan to receive all 6 injections of Radium Ra 223 Dichloride and daily Enzalutamide during the study, per protocol.
7. Subject has received previous strontium-89, samarium-153, rhenium-186, or rhenium-188 for the treatment of bone metastasis within 24 weeks prior to enrollment (Cycle 1/Week 1/Day 1).
8. Subject has received denosumab or Zolendronic Acid for less than 90 days prior to enrollment (Cycle 1/Week 1/Day 1), or if the subject plans to discontinue an anti-resorptive prior to the End of Treatment visit or the last Long Term Follow Up visit.
9. Subject has received an investigational product or experimental therapy within 4 weeks of enrollment (Cycle 1/Week 1/Day 1), or if initiation of either is planned prior to the End of Treatment visit or the last Long Term Follow Up visit.
10. Subject has had treatment with cytotoxic chemotherapy within 4 weeks or enrollment (Cycle 1/Week 1/Day 1), or planned prior to the End of Treatment visit or the last Long Term Follow Up visit, or failure to recover from adverse events due to cytotoxic chemotherapy administered more than 4 weeks prior to enrollment (Cycle 1/Week 1/Day 1), such as persistent myelosuppression, GI toxicity, or severe fatigue. Ongoing neuropathy is not exclusionary.
11. Subject has a history of severe liver insufficiency (r Child-Pugh class B or C).
12. Subject has a history of a myocardial infarction or cardiac arrhythmia within 6 months prior to enrollment (Cycle 1/Week 1/ Day 1).
13. Subject has a history of previous radiotherapy >25% of bone marrow, including hemibody radiation.
14. Subject has a history of any other malignancy within the previous 5 years. A history of squamous or basal cell carcinoma or low-grade superficial bladder cancer that has been adequately treated at least 12 months prior to enrollment is not exclusionary.
15. Subject has undergone major surgery within 4 weeks prior to enrollment (Cycle 1/Week 1/Day 1).
16. Subject has had a blood transfusion or erythropoietin stimulation agents within 4 weeks of enrollment (Cycle 1/Week 1/Day 1).
17. Subject has known imminent or established spinal cord compression.
18. Subject has a serious concurrent medical condition or psychiatric illness.
19. Subject has a history of other serious illness of medical condition including, but not limited to any uncontrolled infection, congestive heart failure New York Heart Association (NYHA) class III or IV, Crohn's Disease or Ulcerative Colitis, uncontrolled hypertension or Bone Marrow Dysplasia at screening.
20. Subject has a gastrointestinal disorder affecting absorption (e.g. gastrectomy, active peptic ulcer disease within 90 days prior to enrollment (Cycle 1/Week 1/Day 1)
21. Subject is not able to swallow the study treatment capsules.
22. Subject has unmanageable fecal incontinence.
23. Subject has any condition that, in the opinion of the investigator, would impair the patient's ability to comply with study procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events and serious adverse events . Adverse events deemed to be related to either study medication will be followed until resolution. | 30 days after the last cycle of Radium Ra 223 dichloride, which will be approximately 7 months after study enrollment

SECONDARY OUTCOMES:
Bone pain measured by the Bone Pain Index- Short Form questionnaire | Thorughout the study and through the last follow-up visit, estimated to be 30 months after study enrollment
  Bone Pain
Quality of Life Questionnaire | Thorughout the study and through the last follow-up visit, estimated to be 30 months after study enrollment
Time to measurable disease progression | Thorughout the study and through the last follow-up visit, estimated to be 30 months after study enrollment
Time to implementation of palliative radiotherapy | Thorughout the study and through the last follow-up visit, estimated to be 30 months after study enrollment
Time to analgesic (Opioid) advancements | Thorughout the study and through the last follow-up visit, estimated to be 30 months after study enrollment
Time from start of Enzalutamide to PSA progression | Thorughout the study and through the last follow-up visit, estimated to be 30 months after study enrollment
Changes and time to total-ALP progression will be measured by recording laboratory values | Thorughout the study and through the last follow-up visit, estimated to be 30 months after study enrollment
  Changes and time to total-ALP progression
Progression to additional antineoplastic therapy will be measured by tracking subject diaries and concomitant medications | Thorughout the study and through the last follow-up visit, estimated to be 30 months after study enrollment
  Progression to additional antineoplastic therapy
Performance status change will be measured by ECOG status | Thorughout the study and through the last follow-up visit, estimated to be 30 months after study enrollment
  Performance status change

CONTACTS AND LOCATIONS:
Overall Officials: Neal D Shore, MD, Principal Investigator — Carolina Research Professionals, LLC
Locations (4):
- United States (4):
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Associated Medical Professionals, Syracuse, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology of Virginia, PLLC, Virginia Beach, Virginia